CLINICAL TRIAL: NCT01514461
Title: A Randomized, Double-blind, Placebo Controlled Study to Assess Efficacy, Safety and Tolerability of LCQ908 in Subjects With Familial Chylomicronemia Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCQ908B2302; 2011-005535-68 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2012-01-23 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Familial Chylomicronemia Syndrome (FCS)
Keywords: Hyperlipoproteinemia (HLP Type I); Fasting Triglycerides
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome; Hyperlipoproteinemias | interventions — pradigastat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- LCQ908 20 mg (Experimental): In period II (0-12 weeks) double-blind treatment: one LCQ908 20 mg active tablet + one LCQ908 placebo matching to 40mg tablet, once daily. No dose titration allowed.
  In period III (12-52 weeks) double blind treatment: Without down titration, the period II dosing regimen will follow. Following decision to down titrate: one LCQ908 10 mg active tablet + one LCQ908 placebo matching to 40 mg tablet + one LCQ908 placebo matching to 10mg tablets, once daily.
  A low fat diet will be followed and recorded in patient diary.
  Interventions: Drug: LCQ908; Drug: Placebo
- LCQ908 40 mg (Experimental): In period II (0-12 weeks) double-blind treatment: one LCQ908 40 mg active tablet + one LCQ908 placebo matching to 20mg tablet, once daily. No dose titration allowed.
  In period III (12-52 weeks) double blind treatment: Without down titration, the period II dosing regimen will follow. Following decision to down titrate: one LCQ908 20 mg active tablet + one LCQ908 placebo matching to 40 mg tablet + one LCQ908 placebo matching to 10mg tablets, once daily.
  A low fat diet will be followed and recorded in patient diary.
  Interventions: Drug: LCQ908; Drug: Placebo
- Placebo (Placebo Comparator): In period II (0-12 weeks) double-blind treatment: one LCQ908 placebo matching to 40mg tablet + one LCQ908 placebo matching to 20mg tablet, once daily.
  In period III (12-52 weeks) double blind treatment: Without down titration, the period II dosing regimen will follow. Following decision to down titrate: one LCQ908 placebo matching to 40mg tablet + one LCQ908 placebo matching to 20mg tablet + one LCQ908 placebo matching to 10mg tablets, once daily.
  A low fat diet will be followed and recorded in patient diary.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCQ908 — LCQ908 10 mg, LCQ908 20 mg, LCQ908 40 mg
  Arms: LCQ908 20 mg; LCQ908 40 mg
Drug: Placebo — LCQ908 10 mg, LCQ908 20 mg, LCQ908 40 mg
  Other Names: LCQ908

SUMMARY:
The purpose of this study is to determine whether LCQ908 is effective and safe in lowering triglycerides in subjects with Familial Chylomicronemia Syndrome (FCS) (Hyperlipoproteinemia [HLP] type I). Data from this study will be used to support a registration submission of LCQ908 20 mg and 40 mg as treatment of chylomicronemia in subjects with FCS (HLP Type 1).

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent given before any assessment was performed for Period I.
2. Male and female patients ages at least 18 years of age.
3. Fasting triglyceride ≥ 8.4 mmol/L (750 mg/dL) at Screening.
4. An established diagnosis of FCS (HLP Type I) confirmed through ultracentrifugation or by documented medical history of a fasting triglyceride ≥ 8.4 mmol/L (750 mg/dL) and by documentation of any of the following at Screening or during the Screening Period:

   * Confirmed homozygote or compound heterozygote for known loss-of-function mutations in Type I-causing genes (such as LPL, apo C II, GPIHBP1, or LMF1)
   * Post heparin plasma LPL activity of ≤ 20% of normal
   * Confirmed presence of LPL inactivating antibodies
5. History of pancreatitis.

Key Exclusion Criteria:

1. Current pancreatitis, pancreatitis was required to be inactive for at least 1 week prior to the screening Visit.
2. Treatment with fish oil preparations within 4 weeks prior to randomization.
3. Treatment with bile acid binding resins (i.e., colesevelam, etc.) within 4 weeks prior to randomization.
4. Treatment with fibrates within 4 weeks prior to randomization.
5. Glybera [alipogene tiparvovec (AAV1-LPLS447X)] gene therapy exposure within the two years prior to screening.
6. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
7. Any surgical or medical conditions, acute or unstable chronic disease which may, based on the investigator's opinion, jeopardize the patient in case of participation in the study or might significantly alter the absorption, distribution, metabolism or excretion of the study drug.
8. History of drug or alcohol abuse within the 12 months prior to randomization or evidence of such abuse at screening.
9. Evidence of liver disease or liver injury as indicated by abnormal liver function tests such as aspartate aminotransferase (AST) and alanine aminotransferase (ALT), or serum bilirubin.
10. Estimated glomerular filtration rate (eGFR) <30mL/min/1.73m2 or history of chronic renal disease.
11. Participation in any clinical investigation within four (4) weeks prior to initial dosing or longer if required by local regulations, or any other limitation of participation based on local regulations.
12. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
13. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive HCG laboratory test.
14. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 100 days after discontinuation of investigational study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Novartis Investigative Site, Seatlle, Washington, United States
- Canada (3):
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Ouest-Montreal
- France (3):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Hamburg
- Novartis Investigative Site, Meibergdreef 9, Netherlands
- Novartis Investigative Site, Cape Town, South Africa
- Spain (2):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
- Novartis Investigative Site, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: In period II (0-12 weeks) double-blind treatment: one LCQ908 placebo matching to 40mg tablet + one LCQ908 placebo matching to 20mg tablet, once daily. In period III (12-52 weeks) double blind treatment: Without down titration, the period II dosing regimen was followed. Following decision to down titrate: one LCQ908 placebo matching to 40mg tablet + one LCQ908 placebo matching to 20mg tablet + one LCQ908 placebo matching to 10mg tablets, once daily. A low fat diet was followed and recorded in patient diary.
- LCQ908 20 mg: In period II (0-12 weeks) double-blind treatment: one LCQ908 20 mg active tablet + one LCQ908 placebo matching to 40mg tablet, once daily. No dose titration allowed. In period III (12-52 weeks) double blind treatment: Without down titration, the period II dosing regimen was followed. Following decision to down titrate: one LCQ908 10 mg active tablet + one LCQ908 placebo matching to 40 mg tablet + one LCQ908 placebo matching to 10mg tablets, once daily. A low fat diet was followed and recorded in patient diary.
- LCQ908 40 mg: In period II (0-12 weeks) double-blind treatment: one LCQ908 40 mg active tablet + one LCQ908 placebo matching to 20mg tablet, once daily. No dose titration allowed. In period III (12-52 weeks) double blind treatment: Without down titration, the period II dosing regimen was followed. Following decision to down titrate: one LCQ908 20 mg active tablet + one LCQ908 placebo matching to 40 mg tablet + one LCQ908 placebo matching to 10mg tablets, once daily. A low fat diet was followed and recorded in patient diary.
Period: Overall Study
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Started | 15 | 15 | 15
Completed | 10 | 12 | 11
Not Completed | 5 | 3 | 4
Not completed — Adverse Event | 2 | 1 | 3
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Patient/guardian decision | 1 | 1 | 1
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (10.9) | 42.3 (13.61) | 42.7 (10.94) | 45.9 (12.63)
Age, Customized [Number; unit: Participants]
  < 65 years | 12 | 15 | 15 | 42
  >=65 years | 3 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 4 | 19
  Male | 7 | 8 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Fasting Triglycerides From Baseline to 12 Weeks
Description: Blood samples were collected for a fasting lipid panel, including triglycerides. If the 12-week value was missing, the measurement value at 12 weeks or the last available post-baseline measurement value during the double-blind treatment period was analyzed. Baseline is defined as the average of fasting triglyceride values taken at day -3 and day 1. Adjusted geometric means are calculated by back-transforming the adjusted means from the model and expressing as a percentage change from baseline.
Time Frame: Baseline to 12 weeks
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized. The number of randomized patients with non-missing fasting triglycerides values at baseline and Week 12 are included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Groups:
- LCQ908 20mg: In period II (0-12 weeks) double-blind treatment: one LCQ908 20 mg active tablet + one LCQ908 placebo matching to 40mg tablet, once daily. No dose titration allowed. In period III (12-52 weeks) double blind treatment: Without down titration, the period II dosing regimen was followed. Following decision to down titrate: one LCQ908 10 mg active tablet + one LCQ908 placebo matching to 40 mg tablet + one LCQ908 placebo matching to 10mg tablets, once daily. A low fat diet was followed and recorded in patient diary.
Arm/Group | Placebo | LCQ908 20mg | LCQ908 40 mg
Number analyzed (Participants) | 14 | 14 | 12
percent change | 45.6 [6.8 to 98.7] | 3.7 [-24.3 to 42.1] | -13.9 [-38.9 to 21.3]
Statistical Analysis 1: Comparison: Placebo vs LCQ908 20mg; Test type: Superiority or Other; p = 0.0538, Mixed Models Analysis; Mixed Model of Repeated Measurements; % change from reference treatment = -28.78, 95% CI 2-sided [-55.69 to 14.46]
Statistical Analysis 2: Comparison: Placebo vs LCQ908 40 mg; Test type: Superiority or Other; p = 0.0182, Mixed Models Analysis; Mixed Model of Repeated Measurements; % change from reference treatment = -40.88, 95% CI 2-sided [-63.99 to -2.94]

2. Secondary Outcome: Percentage of Patients Responding to Investigational Treatment by Achieving Fasting Triglycerides (TG) of at Least 40% From Baseline or Final Fasting TG < 8.4 mmol/L (750 mg/dL)
Description: Percentage calculated as (m/n)*100 where m = number of patients who respond; n = the number of patients with non-missing fasting triglyceride.
Time Frame: Baseline, 12 weeks, 24 weeks, 52 weeks
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 15 | 15 | 15
Percentage of participants
  Week 12 (n = 14, 14, 12) | 14.3 | 21.4 | 50.0
  Week 24 (n = 13, 14, 12) | 30.8 | 35.7 | 33.3
  Week 52 (n = 11, 14, 11) | 18.2 | 21.4 | 27.3

3. Secondary Outcome: Percentage of Patients Responding to Investigational Treatment by Achieving Final Fasting Triglycerides < 8.4 mmol/L (750 mg/dL)
Description: as for outcome 2
Time Frame: 12 weeks, 24 weeks, 52 weeks
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 15 | 15 | 15
Percentage of participants
  Week 12 (n = 14, 14, 12) | 14.3 | 14.3 | 33.3
  Week 24 (n = 13, 14, 12) | 30.8 | 14.3 | 16.7
  Week 52 (n = 11, 14, 11) | 18.2 | 14.3 | 18.2

4. Secondary Outcome: Percentage of Patients Responding to Investigational Treatment by Achieving Fasting Triglycerides (TG) of at Least 40% From Baseline
Description: as for outcome 2
Time Frame: Baseline, 12 weeks, 24 weeks, 52 weeks
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 15 | 15 | 15
Percentage of participants
  Week 12 (n = 14, 14, 12) | 0.0 | 14.3 | 25.0
  Week 24 (n = 13, 14, 12) | 15.4 | 28.6 | 16.7
  Week 52 (n = 11, 14, 11) | 0.0 | 14.3 | 27.3

5. Secondary Outcome: Percentage of Patients Achieving Fasting Triglycerides (TG) Target Thresholds
Description: Percentage of patients reaching target values of <1000 mg/dL or target values of < 2000 mg/dL for fasting triglycerides is reported. Pecentage calculated as (m/n)*100; where 'm' The number of patients who reach target values for fasting triglyceride, 'n' the number of patients with non-missing fasting triglyceride.
Time Frame: 12 weeks, 24 weeks, 52 weeks
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized.
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 15 | 15 | 15
Percentage of patients
  TG < 1000 mg/dL, week 12 (n=14,14,12) | 14.3 | 21.4 | 33.3
  TG < 1000 mg/dL, week 24 (n=13,14,12) | 30.8 | 21.4 | 25.0
  TG < 1000 mg/dL, week 52 (n=11,14,11) | 27.3 | 14.3 | 36.4
  TG < 2000 mg/dL, week 12 (n=14,14,12) | 35.7 | 50.0 | 83.3
  TG < 2000 mg/dL, week 24 (n=13,14,12) | 38.5 | 57.1 | 58.3
  TG < 2000 mg/dL, week 52 (n=11,14,11) | 36.4 | 50.0 | 63.6

6. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides
Time Frame: Baseline, 24 weeks, 52 weeks
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 15 | 15 | 15
Percent change
  Week 24 (n=13, 14, 12) | 4.9 [-26.6 to 50.1] | -15.8 [-40.5 to 19.3] | 5.5 [-28.0 to 54.5]
  Week 52 (n=11, 14, 11) | 15.2 [-23.0 to 72.5] | -6.7 [-36.4 to 36.9] | 4.9 [-31.2 to 60.0]

7. Secondary Outcome: Percent Change From Baseline for Postprandial Triglycerides Following the Standardized Meal Tolerance Test at Week 12
Description: Post prandial peak triglycerides - maximum triglyceride value over 0-24 hours Post prandial triglycerides AUC0-24 - area under the time curve for triglycerides over 0-24 Adjusted geometric means are calculated by back-transforming the adjusted means from the model and expressed as a percentage change from baseline. hours
Time Frame: 0-24 hours at Baseline, Week 12
Population: Full analysis set (FAS) consisted of all randomized patients, except for those who were mis-randomized. For each category, the number of randomized patients who have non-missing values are included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 15 | 15 | 15
Percent change
  Triglycerides (Peak 0-24h) [n=12, 12, 11) | 56.9 [6.9 to 130.2] | 8.6 [-24.8 to 56.8] | 6.3 [-30.3 to 62.2]
  Triglycerides (AUC 0-24h) [n=12, 12, 11) | 44.5 [-1.3 to 111.5] | 0.8 [-30.1 to 45.1] | 2.8 [-32.4 to 56.3]

8. Secondary Outcome: Pharmacokinetics of LCQ908 - Trough Concentration (Cmin) and Observed Maximum Blood Concentration (Cmax)
Description: Lowest observed blood concentration (Cmin) and observed maximum blood concentration (Cmax) following drug administration derived from non-compartmental analysis using scheduled sampling time for the whole dataset.
Time Frame: 0, 1, 2, 3, 4, 6, and 24 hours at Week 12
Population: Safety set (SAF) consisted of all patients who received at least one dose of study drug and had at least one post-baseline safety assessment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 12 | 9
ng/mL
  Cmin | 312 (120) | 426 (224)
  Cmax | 603 (244) | 745 (408)

9. Secondary Outcome: Pharmacokinetics of LCQ908- Area Under the Plasma Concentration Time Curve AUC (0-24hour)
Description: The area under the concentration-time curve from time zero to 24 hours after drug administration was calculated by using linear trapezoidal rule.
Time Frame: 0, 1, 2, 3, 4, 6, and 24 hours at Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL *hr
Arm/Group | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 12 | 9
ng/mL *hr | 11000 (4100) | 14300 (7390)

10. Secondary Outcome: Pharmacokinetics of LCQ908- Time to Reach Maximum Concentration Following Drug Administration Tmax (Hours)
Time Frame: 0, 1, 2, 3, 4, 6, and 24 hours at Week 12
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 12 | 9
hours | 6 [0 to 24] | 8 [0 to 24]

11. Secondary Outcome: Pharmacokinetics of LCQ908- Average Observed Blood Concentration (Cavg)
Description: Average observed blood concentration measured by (AUC0-24)/24.
Time Frame: 0, 1, 2, 3, 4, 6, and 24 hours at Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 12 | 9
ng/mL | 459 (171) | 597 (308)

12. Secondary Outcome: Number of Patients Reported With Any Adverse Event, Serious Adverse Event and Death
Time Frame: 52 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Number analyzed (Participants) | 15 | 15 | 14
Participants
  At least one adverse events | 15 | 15 | 14
  At least one serious adverse event | 6 | 6 | 3
  Death | 1 | 0 | 0

ADVERSE EVENTS:
Description: Safety set (SAF) consisted of all patients who received at least one dose of study drug and had at least one post-baseline safety assessment.
Arm/Group | Placebo | LCQ908 20 mg | LCQ908 40 mg
Serious Adverse Events (participants affected / at risk) | 6/15 | 6/15 | 3/14
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | LCQ908 20 mg (N=15) | LCQ908 40 mg (N=14)
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 2 | 3 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 | 2 | 1
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
MALIGNANT PALATE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | LCQ908 20 mg (N=15) | LCQ908 40 mg (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 0 | 1
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0 | 0
DEAFNESS (Ear and labyrinth disorders) | 0 | 1 | 0
BLEPHARITIS (Eye disorders) | 0 | 1 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 7 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 1
ABDOMINAL RIGIDITY (Gastrointestinal disorders) | 0 | 0 | 1
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 0 | 1 | 0
CHANGE OF BOWEL HABIT (Gastrointestinal disorders) | 1 | 2 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 0
DEFAECATION URGENCY (Gastrointestinal disorders) | 1 | 0 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 10 | 12 | 10
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 2 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 1 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1 | 0
FAECES SOFT (Gastrointestinal disorders) | 0 | 1 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 1 | 1
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 0 | 0
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 5 | 4
PANCREATITIS (Gastrointestinal disorders) | 0 | 3 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 6 | 4
ASTHENIA (General disorders) | 0 | 1 | 2
CYST (General disorders) | 1 | 1 | 0
FATIGUE (General disorders) | 2 | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 1 | 2 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 0 | 1 | 0
ALLERGY TO PLANTS (Immune system disorders) | 1 | 0 | 0
FOOD ALLERGY (Immune system disorders) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 1
CONJUNCTIVITIS (Infections and infestations) | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 1 | 0 | 0
EAR INFECTION (Infections and infestations) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 3 | 2 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 0
HAND-FOOT-AND-MOUTH DISEASE (Infections and infestations) | 0 | 0 | 1
HORDEOLUM (Infections and infestations) | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 3 | 0 | 4
JOINT ABSCESS (Infections and infestations) | 1 | 0 | 0
LARYNGITIS (Infections and infestations) | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 2 | 4
PHARYNGITIS (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
RHINITIS (Infections and infestations) | 0 | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0 | 0
TINEA INFECTION (Infections and infestations) | 0 | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
CHEST INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
SCAR (Injury, poisoning and procedural complications) | 1 | 0 | 0
SPORTS INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 1
CAROTID BRUIT (Investigations) | 1 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 0 | 2 | 2
WEIGHT INCREASED (Investigations) | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 2 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCLE FATIGUE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
NEOPLASM SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 3 | 3 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 1
HEADACHE (Nervous system disorders) | 1 | 4 | 1
LETHARGY (Nervous system disorders) | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 2 | 1
SYNCOPE (Nervous system disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 2 | 0 | 0
STRESS (Psychiatric disorders) | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ROSACEA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
XANTHOMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
HOT FLUSH (Vascular disorders) | 0 | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.